CLINICAL TRIAL: NCT02474277
Title: How Well Does the 30-second Chair Stand Test Predict Rehabilitation Needs in Acutely Admitted Elderly Patients?
Brief Title: How Well Does the 30-Second Chair Stand Test Predict Rehabilitation Needs in Acutely Admitted Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Christian Backer Mogensen, Ass. professor, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SLB-ED-08-2014
Record Dates: First submitted 2014-12-10; First posted 2015-06-17 (Estimated); Last update posted 2015-06-17 (Estimated); Status verified 2015-06

CONDITIONS: Acute Disease
MeSH Terms: conditions — Acute Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 30 sec chair stand test (Other): all patients in this Group receives a diagnostic test for functional impairment
  Interventions: Other: 30 sec chair stand test

INTERVENTIONS:
Other: 30 sec chair stand test — diagnostic test for functional impairment

SUMMARY:
The aims are to identify predictive indicators of hospitalized elderly medical patients' need for rehabilitation and to validate (known group validity) the Chair Stand Test

DETAILED DESCRIPTION:
In the emergency department the assessment of acutely admitted elderly medical patients' need for rehabilitation is difficult as it has to been performed within 48 hours. Is it possible to use the the Chair Stand Test in combination with admission complaints and identified risk factors to predict the need for rehabilitation? An investigating of the Chair Stand Test is needed, as its validity with hospitalized patients is undocumented.

ELIGIBILITY:
Inclusion Criteria:

* Can speak and understand Danish
* Can report personal data
* Within the first 48 hours of admission are able to sin on an ordinary chair

Exclusion Criteria:

* Patients ordinarily unable to walk

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 156 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
30-Second Chair Stand Test | 14 days after admission at the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Christian B Mogensen, MD PHD, Principal Investigator — University of Southern Denmark
Locations (1):
- Lillebaelt hospital, Kolding, Kolding, Denmark

REFERENCES:
- [Derived] Bruun IH, Maribo T, Norgaard B, Schiottz-Christensen B, Mogensen CB. A prediction model to identify hospitalised, older adults with reduced physical performance. BMC Geriatr. 2017 Dec 7;17(1):281. doi: 10.1186/s12877-017-0671-5. PMID 29216838